CLINICAL TRIAL: NCT06528158
Title: Sibling Group for Children and Teenagers Living with a Sibling Who Suffers from Anorexia Nervosa: a Pilot Acceptability Study
Brief Title: Speech Groups for Children Living with a Sibling Who Suffers from Anorexia Nervosa
Acronym: EMA-FRaM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0181
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: siblings; groups; children; teenagers; acceptability
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: sibling group — The group will be based on a systemic model and led by two child psychiatrists trained in family and multi-family therapy, who will not subsequently be involved in the data analysis. It will consist of 4 sessions of 1h30, spread over a period of 2 months, with a maximum of 8 participants per session. The first 3 sessions will be spaced 15 days apart, and the last session will take place 3 weeks apart from the third session.
  The characteristics of the group (frequency, duration, number of sessions and participants) were built on data from the literature as well as on clinical feedback from a first pilot group conducted in January and February 2024 on the Toulouse pediatric unit by the two therapists who will lead the groups during the study.

SUMMARY:
Anorexia nervosa (AN) is a complex mental disease with a huge impact on the patient's siblings life and well-being. Based on literature, group interventions for siblings of children suffering from a chronic disease could provide an effective support. A few have been studied, and even fewer exist for siblings of children with AN.

DETAILED DESCRIPTION:
AN has a significant impact on nuclear family (parents and siblings). An emerging literature highlights the need for a particular attention to siblings. Despite this evidence, research and clinical applications still lack in this area. Indeed, most of health services in AN offer support for patients, family, parents, but only few specific support for siblings, although positive outcomes of sibling group interventions were reported in other somatic and psychic disabilities.

Noting the gap between the need and the lack of specific support, the study hypothesis is that the poor diffusion of these interventions in AN might result from a low acceptability. The study propose to explore acceptability to adapt and improve group intervention for siblings of children and teenagers receiving care for anorexia nervosa.

The study is a mixed-method pilot study assessing the acceptability of a group intervention by including a maximum of 24 siblings of children suffering from AN, aged from 8 to 18, across three group sessions, each consisting of 4 meetings. All participants will be invited to fulfill two different auto-questionnaires about their quality of life (before and after group session) and the intervention's acceptability (after group session).

Quantitative data will be complemented with qualitative data, collected from individual semi-structured interviews with a targeted sampling among group participants.

ELIGIBILITY:
* inclusion criteria : Sibling presenting a DSM (Diagnostic and Statistical Manual)-5 of Mental Disorders diagnosis of AN, and engaged in inpatient or outpatient healthcare
* exclusion criteria :

  * (1) Opposition from the participant and/or from their legal representatives.
  * (2) Non-fluent French speaker
  * (3) Clinical presentation not compatible with the group sessions

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Maximum 24 participants will overall be included to attend group sessions. Around 15 participants will be invited to an individual interview after group sessions.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Group ACCEPTABILITY | after attending group sessions, maximum 3 months after baseline
  assess the clinical setting " sibling group "'s acceptability among siblings of teenagers engaged in health care for AN. This will be assessed through the acceptability scale Abbreviated Acceptability Rating Profile (AARP) after attending group sessions.
  In the questionnaire, there are 8 questions. For each, a scale of 1 to 6, with 1 being "not agreeing at all with the question" and 6 being "completely agree". Maximum score = 48 the higher the score, the better the acceptability of the group is felt by participants.

SECONDARY OUTCOMES:
Impact of the groups on quality of life | baseline
  THE PEDIATRIC QUALITY OF LIFE INVENTORY VERSION 4 (PEDSQLTM4.0) (MODULE GENERIC CORE SCALE) The PedsQL is a modular instrument for measuring health-related quality of life (HRQOL) in children and adolescents ages 2 to 18.
  The PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent proxy-report scales developed as the generic core measure to be integrated with the PedsQL Disease-Specific Modules.
  The PedsQL 4.0 Generic Core Scales consist of 23 items A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is us
impact of the groups on quality of life | after attending group sessions, maximum 3 months after baseline
  THE PEDIATRIC QUALITY OF LIFE INVENTORY VERSION 4 (PEDSQLTM4.0) (MODULE GENERIC CORE SCALE) The PedsQL is a modular instrument for measuring health-related quality of life (HRQOL) in children and adolescents ages 2 to 18.
  The PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent proxy-report scales developed as the generic core measure to be integrated with the PedsQL Disease-Specific Modules.
  The PedsQL 4.0 Generic Core Scales consist of 23 items A 5-point response scale is used across the child self-report (for ages 8 to 18) and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). A 3-point scale is us

CONTACTS AND LOCATIONS:
Overall Officials: Antoine STOCKER, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UH Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No